CLINICAL TRIAL: NCT06113783
Title: A Post-market, Randomized, Controlled Clinical Investigation to Assess the Efficacy of HYALUBRIX 60® Intra-articular Injection in the Symptomatic Relief of Knee Osteoarthritis
Brief Title: Assessment of Efficacy of a Single Intra-articular Injection of HYALUBRIX 60 in Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fidia Farmaceutici s.p.a. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EQB7-20-02
Record Dates: First submitted 2023-10-30; First posted 2023-11-02 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2023-10

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: post-market, monocentre, randomized, controlled clinical investigation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1- ACTIVE (Experimental): Intra-articular injection at baseline of HYALUBRIX 60® plus PEP 3 times a week at home for the 12 months of observation;
  Interventions: Device: HYALUBRIX 60
- Group 2-CONTROL (No Intervention): Physical Exercise Program alone 3 times a week at home for the 12 months of observation.

INTERVENTIONS:
Device: HYALUBRIX 60 — 1.5% solution of non-modified HA (60mg/4ml) obtained from bacterial fermentation with high molecular weight.
  Other Names: HYALONE
  Arms: Group 1- ACTIVE

SUMMARY:
The purpose of this study is to evaluate the effect of one single intra-articular (IA) injection of HYALUBRIX 60® plus physical exercise program (PEP) in terms of pain reduction, compared to PEP alone, in patients with knee osteoarthritis (OA).

DETAILED DESCRIPTION:
Knee Osteoarthritis (OA) is one of the primary causes of pain and disability worldwide, associated with functional restrictions, morphological changes in the subchondral bone, articular cartilage degeneration and damage to the surrounding soft tissue. [Heiden TL, 2009; Di Cesare PE, 2009, Fernandes L, 2013].

In the degradation of articular cartilage, functional limitation and pain, underlies the quantitative and qualitative alteration of hyaluronic acid (HA), the main component of synovial fluid and cartilage, in a pathophysiological process influenced by a wide variety of risk factors [Balazs, E.A, 1993]. In OA patients, HA is depolymerized and eliminated faster than in healthy subjects, due to chronic inflammation [Legré-Boyer, V., 2015]. HA concentration is significantly decreased in patients with end-stage knee OA [Bagga, H et al, 2006].

HA used intra-articularly in the treatment of OA is known to increase viscosity of the synovial fluid, facilitate gliding via layer formation on the cartilage and protect soft tissue from trauma by acting as a shock absorbent [Legré-Boyer et al., 2015; Cooper et al., 2017; Bowman et al., 2018]. HA also soothes the pain and exerts an immunomodulatory effect on inflammatory cells [Pelletier, J.P, 1993]. HA has a delayed onset of action in comparison with IA corticosteroids, but a longer-lasting benefit [Bannuru, R.R., 2009].

HYALUBRIX 60® is a CE-marked medical device of class III consisting in a 1.5% solution of non-modified HA (60mg/4ml) obtained from bacterial fermentation with high molecular weight. HYALUBRIX 60® exhibits a behavior very similar to the synovial fluid that it replaces. In particular, it confers proper rheological properties, trans-synovial fluid buffering, and permeability to metabolites and macromolecules.

This post-market, monocentre, randomized, controlled clinical investigation is designed to enrol a relatively young, active population of subjects with knee OA and to compare responses to treatment with one IA HYALUBRIX 60® injection plus physical exercise program (PEP), versus a PEP alone. Because PEP or exercise programs may be considered the first line standard of care in OA knee pain, particularly in younger, active patients [Nelson AE et al. 2014], the hypothesis of the study is that HYALUBRIX 60® combined to PEP, provides greater relief of pain associated with knee OA in the enrolled study subjects than with use of PEP alone. The primary endpoint pain relief is measured after 2 months, but observation will last up to 12 months and effects on both pain relief and physical function will be evaluated at 1, 2, 6, and 12 months after single injection (in the HYALUBRIX 60® treated arm), through WOMAC index.

Selection of dose was done on the basis of a previous randomised clinical trial (RCT) (Clementi et al, 2018) conducted on 50 patients, that showed no significant difference between the two groups (single injection and injection repeated after 3-4 weeks) for beneficial long-term pain relief and functional improvement in terms of VAS score, WOMAC score and Lequesne index at 1, 3, 6 and 12 months. A clinical improvement was observed as early as at 1 month in each treatment group and continued until 1 year with no difference in the development over time between the two treatment groups.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily given informed consent to investigation participation in writing encompassing consent to data recording and verification procedures;
2. Male or female subjects aged ≥18 years and ≤70 years with active life-style;
3. BMI ≤40 kg/m2;
4. Patients affected by knee osteoarthritis, as defined by American College of Rheumatology (ACR) clinical and radiographic criteria for OA of the knee, and meeting the following conditions:

   * Kellgren-Lawrence Grade 2 to 3 severity OA of the target knee with presence of osteophytes determined from X-rays of the knee obtained within 6 months from the screening visit; i.e. in the tibio-femoral compartment of the target knee with at least 1 osteophyte and measurable joint space, as diagnosed by standard X-rays (anterior- posterior view [weight bearing extension or semi-flexion] and lateral). In the case that a patient has not a valid X-ray within 6 months prior to screening, the exam is to be performed during the screening period;
   * Patients suffering from OA symptoms of the target knee for at least 3 months prior to the screening visit; Note: patients with bilateral OA of the knee will be allowed as long as they can differentiate pain in the target knee, do not need to use analgesics for treatment of their contralateral knee, and do not expect to receive treatment of the contralateral knee during the investigation. In the case that both knees are eligible for the investigation based on pain intensity, the knee with the greater pain VAS score on the WOMAC pain VAS A1 subscale (walking on a flat surface) will be selected as the target knee;
5. Pain ≥50 mm on the WOMAC pain VAS A1 subscale (walking on a flat surface) in the target knee;
6. Patients having discontinued use of all systemic analgesic/non-steroidal anti-inflammatory drugs (NSAIDs) therapy for at least 7 days (24 hours for paracetamol) prior to the screening visit and agree not to resume them during the investigation. Note: paracetamol will be provided to patients as rescue medication.
7. If female of child-bearing potential, must have a negative urine pregnancy test at the screening visit and use a reliable form of contraception for more than 1 month prior to Screening and throughout the investigation. Note: to be considered females of non-child- bearing potential, females must be surgically sterile or postmenopausal as documented in medical history for at least 1 year. Highly effective birth control methods include: combined hormonal contraception (containing estrogens and progestogen) associated with inhibition of ovulation (oral, intravaginal, transdermal); progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable); intrauterine device (IUD); intrauterine hormone-releasing system (IUS); bilateral tubal occlusion; vasectomised partner; sexual abstinence.*

   * Note: According to 4.1 paragraph "Birth control methods which may be considered as highly effective" of the Clinical Trial Facilitation Group (CTFG)/Recommendations related to contraception and pregnancy testing in clinical trials.

Exclusion Criteria:

1. Radiographic assessment confirming abnormal patellofemoral tracking or articulation or abnormal/excessive patellar subluxation in lateral view;
2. Major injury to or disorder of the contralateral knee or other weight-bearing joint that would interfere with the study assessments;
3. Secondary OA due to a prior or concomitant condition (e.g., septic arthritis, inflammatory joint disease, gout, articular fracture, major dysplasia, or congenital abnormality, hemochromatosis, etc.);
4. Patients who have had arthroplasty at the target knee at any time;
5. Surgery in the target knee within the previous 12 months prior to Screening or any planned surgery throughout the duration of the investigation;
6. Surgery in the contralateral knee or other weight-bearing joint within the previous 12 months that would interfere with the study assessments;
7. Patients that are candidate for knee replacement within the next 12 months;
8. Patients having had diagnostic or surgical knee arthroscopy, or knee lavage in the target knee in the 6 months prior to the screening visit, or patients in which such procedures are planned during the study;
9. Patients with total joint replacement implants, unicondylar implants or patellofemoral replacement implants in the study joint;
10. Ligament reconstruction of the target knee in the previous 3 years;
11. Inflammatory arthropathies such as rheumatoid arthritis, lupus, or psoriatic arthritis;
12. Patients with clinically relevant intra-articular effusion of the target knee;
13. Episode of gout or calcium pyrophosphate (pseudogout) diseases within 6 months prior to Screening;
14. Patients having received:

    * Corticosteroids by systemic administration within 30 days prior to the screening visit.

    Inhaled corticosteroids are permitted if the Subject has been on a stable regimen for the past 1 month prior to Screening and remains on this regimen throughout the course of the investigation;
    * Analgesic/NSAIDs by systemic administration within 7 days prior to the screening visit;
    * Intra-articular drugs within 12 weeks prior to the screening visit;
    * Chondroitinsulphate, glucosamine, diacereine, bisphosphonates or matrix metalloproteinase (MMP) inhibitors within 30 days prior to the screening visit;
    * Viscosupplementation of the target knee within 6 months prior to the screening visit;
    * Paracetamol in the 24 hours prior to the screening visit;
    * Treatment with any other investigational product within 3 months prior to the screening visit.
15. History of allergic reaction to an intra-articular Hyaluronic acid injection;
16. Known hypersensitivity (allergy) to gram positive bacterial proteins;
17. Inability to perform the Timed Up and Go (TUG) test;
18. X-ray findings of acute fractures, severe loss of bone density, avascular necrosis and/or severe deformity;
19. Axial deviation of the lower limbs greater than 20 degrees in valgus or varus on standing X-ray, ligamentous laxity, or meniscal instability as per study investigator(s);
20. Significant surgery of lower limbs (hip, ankle, foot) that may interfere with knee assessments;
21. Patients with any musculoskeletal condition affecting the target knee that would impair assessment of the effectiveness in the target knee (e.g. Paget's disease of bone);
22. Patients with significant pain outside the target knee, including significant hip or back pain;
23. Chronic use of analgesia for pain (including pain in the other knee or any other joint) that may interfere with the evaluations of the test knee (such as possible use of rescue medication for these other conditions);
24. Known allergies to paracetamol and hyaluronan preparations;
25. Recurrent medical history of severe allergic or immune-mediated reactions;
26. Active infection or skin diseases in the area of the potential injection site or joint;
27. Any dermatological disease overlying the study joint that would contraindicate injections or aspirations;
28. Peripheral neuropathy that would be severe enough to interfere with the evaluation of the subject;
29. Psychological status (e.g., anxiety, depression, poor sleep quality, pain catastrophizing, etc.) that may interfere with functional assessment of the target knee;
30. Vascular insufficiency of lower limbs that is severe enough to interfere with the evaluation of the subject;
31. Any concomitant disease(s) or condition(s) that may interfere with the free use and evaluation of the affected knee for the 12 months course of the investigation (cancer, other rheumatic diseases, gout, severe congenital defects, etc.);
32. Continued participation in an experimental drug/device study or any clinical trial within the previous 8 weeks prior to Screening. Subjects must have fully completed participation in an experimental drug/device study of any clinical trial at least 8 weeks prior to screening;
33. Pregnancy, breastfeeding, planned conception, premenopausal women who have not had tubal ligation, hysterectomy, or are unwilling or unable to utilize contraceptive measures (or contraception);
34. Prior history of any malignancy with the exception of basal cell carcinoma of the skin treated more than 2 years prior to Screening;
35. Significant bleeding diathesis;
36. Patients who are not able to comply with study procedures or who are likely to be noncompliant or uncooperative during the study according to the investigator's opinion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-16 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Pain reduction from baseline | 2 months
  Pain intensity will be measured by means of the WOMAC Pain VAS scale (Scale A) (1-100 mm). The mean change in WOMAC Pain VAS score in the target knee from baseline to 2 months will be the primary efficacy endpoint.

SECONDARY OUTCOMES:
Pain reduction from baseline | 1,2, 6 and 12 months
  Pain intensity will be measured by means of the WOMAC Pain VAS scale (Scale A) (1-100 mm). The mean change in WOMAC Pain VAS score in the target knee
Reduction of Stiffness, physical function and overall WOMAC in the target knee from baseline | 1,2, 6 and 12 months
  Stiffness, physical function and overall WOMAC improvement, as change of WOMAC scores (Scale B, C, Total WOMAC) (1-100 mm) in the target knee
Treatment response from baseline | 1, 2, 6 and 12 months
  Change in WOMAC Pain, Physical Function and Stiffness subscale in the target knee of 0-30%, 31-50%, 51-70%, 71-90%, >90% or worsening from baseline
EQ-5D-5L score changes from baseline | 2, 6, 12 months
  EQ-5D is a general, preference-weighted health status instrument that asks patient questions about their overall health status and Health-Related Quality of Life (HRQoL). EQ-5D measures health status using the following 5 dimensions: mobility, self-care, usual activity, pain/discomfort, and anxiety/depression. EQ-5D has 3L and 5L versions, and 5L could increase the reliability and sensitivity (discriminatory power) while feasibility and potentially reducing ceiling effects, compared with 3L. EQ-5D-5L includes 5 levels of severity in each of five dimensions: no problem, slight problems, moderate problems, severe problems, and extreme problems.
Improvement of physical function from baseline | 2, 6, 12 months
  Improvement of physical function such as strength, balance, and agility as differences of Time Up to Go (TUG) test performance from baseline to 1, 2, 6 and 12 months. The TUG is a transition test that assesses strength, agility and dynamic balance during multiple activities including sit-to-stand, walking short distances and changing direction whilst walking. The TUG measures (in seconds) the time taken to stand up from a standard armchair (approximate seat height of 46 cm, arm height of 65 cm), walk a distance of 3m, turn around, walk back to the chair and sit down.
Rescue medication (paracetamol) daily consumption from baseline | 12 months
  The consumption of daily rescue medication (paracetamol) in the overall study period required for pain relief will be evaluated using a patient diary. The number and percentage of patients who will take at least one dose of rescue medication, as well as the total amount of rescue medication taken over the study, will be analyzed.
Number of subjects that switched to HYALUBRIX 60® Group due to PEP failure | 2 months
  The study provides for subjects randomized to the PEP alone study group to cross over to HYALUBRIX 60® if improvement has not been achieved by the 2-month follow up visit.
Number of Adverse Events related to the treatment | 12 months
  Safety of HYALUBRIX 60® will be evaluated in terms of incidence of treatment-emergent adverse events (TEAEs) over the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Valter Santilli, Principal Investigator — UOC Medicina Fisica e Riabilitativa SMC09, AOU Policlinico Umberto I, Rome, Italy
Locations (1):
- UOC Medicina Fisica e Riabilitativa SMC09, AOU Policlinico Umberto I, Rome, Italy, Roma, Italy

IPD SHARING:
Plan to Share IPD: No